CLINICAL TRIAL: NCT01034917
Title: Pilot Study to Assess the Efficacy and Safety of Switching Protease Inhibitor to Etravirine in HIV-1-infected Subjects With Viremia Suppression
Brief Title: Switching From Protease Inhibitor (PI) to Etravirine in HIV-1 Infected Subjects With Viremia Suppression
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Germans Trias i Pujol Hospital (Other)
Responsible Party: Principal Investigator, Dra. EUGENIA NEGREDO PUIGMAL, Dra. Eugenia Negredo Puigmal, Fundación FLS de Lucha Contra el Sida, las Enfermedades Infecciosas y la Promoción de la Salud y la Ciencia
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ETRA-SWITCH
Record Dates: First submitted 2009-12-17; First posted 2009-12-18 (Estimated); Last update posted 2020-01-31 (Actual); Status verified 2020-01

CONDITIONS: HIV
Keywords: Active Comparator; Placebo Comparator; Sham Comparator; No intervention; Other; Treatment Experienced
MeSH Terms: interventions — etravirine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Etravirine group (Experimental): To switch from the PI to Etravirine 400 mg dissolved in water every 24 hours
  Interventions: Drug: Etravirine 400 mg dissolved in water every 24 hours
- Control group (Active Comparator): Continue with the same antiretroviral regimen
  Interventions: Drug: Continue with the same antiretroviral regimen

INTERVENTIONS:
Drug: Etravirine 400 mg dissolved in water every 24 hours — Switch from the PI to Etravirine 400 mg dissolved in water every 24 hours
  Other Names: ETV
  Arms: Etravirine group
Drug: Continue with the same antiretroviral regimen — Continue with the same antiretroviral regimen
  Other Names: CNT
  Arms: Control group

SUMMARY:
This is a 48 week randomized, prospective, controlled, open-label, proof-of-concept pilot clinical trial.

Patients with HIV-1 infection on HAART PI-based regimen will be randomized to switch from the PI to etravirine (400 mg dissolved in water every 24 hours) or to continue with the same approach.

The aim of the study is to compare the virological efficacy of the etravirine-based regimen with standard PI-containing regimen.

DETAILED DESCRIPTION:
Etravirine is a second generation non-nucleoside analogue reverse transcriptase inhibitor (NNRTI) approved by the U.S. Food and Drug Administration (FDA) in January 2008 and by the European Medicines Agency in September 2008 for clinical use in adults with incomplete virologic suppression and resistance to previous NNRTI and other antiretroviral classes.

A question that has not been explored is whether subjects with sustained undetectable HIV-1 RNA-levels experiencing antiretroviral-related toxicity can safely switch their current PI to etravirine. This treatment strategy could allow improvements in tolerability and lipid profile and would permit an easy posology (400 mg dissolved in water every 24 hours). We designed a proof-of-concept study to test the efficacy and safety of switching from a Protease Inhibitor (PI) to etravirine in subjects with viral suppression as an antiretroviral strategy of simplification therapy, based on the high antiviral potency, low toxicity, together with its easy posology (in water dissolution).

Patients with HIV-1 infection on HAART PI-based regimen will be randomized to switch from the PI to etravirine (400 mg dissolved in water every 24 hours) or to continue with the same approach.

The primary endpoint would be the percentage of patients who maintain virological suppression at week 48.

ELIGIBILITY:
Inclusion Criteria:

1. Adult patient having a diagnosis of HIV-1 infection.
2. Antiretroviral therapy started at least 12 months before, always with a HAART combination including 2 NRTIs plus a PI.
3. Maintained undetectable plasma HIV-1 RNA (VL < 50 copies/mL) since the beginning of antiretroviral therapy, for at least 6 months.
4. Absence of suspected or documented resistance mutations in the RT associated to NNRTIs or to any NRTI.
5. Patient having at least one of the following conditions:

   * Dyslipemia (LDL cholesterol >130 mg/dL or triglycerides > 350 mg/dL) derived from their current PI regimen or current use of lipid-lowering agents due to dyslipemia,
   * Antiretroviral-related gastrointestinal disturbances, or
   * Low patient's satisfaction associated with the current regimen posology (BID regimen, ritonavir use, ritonavir intolerance…).
6. Good treatment adherence.
7. Voluntary written informed consent.

Exclusion Criteria:

1. Previous therapy with mono or dual antiretroviral therapies after initial of HAART era.
2. Previous antiretroviral treatment failures, treatment interruptions (A) or blips (B) in viral load (VL > 50 copies/mL).
3. Acute infections or uncontrolled chronic infection in the 2 months previous to the inclusion.
4. Pregnancy or fertile women willing to be pregnant.
5. Clinically significant malabsorption syndrome within 30 days prior to randomization.

(A) Patients who in the past made any interruption of treatment (provide that it has not been in the last year) may be considered candidates for the study, if they meet other criteria for inclusion, since the break in the treatment should not assume the emergence of mutations.

(B) Small blips that are preceded or forwarded by 2 undetectable viral loads will not be taken in care.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 43 (Actual)
Dates: Start 2009-12; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
Viral load | week 48 after baseline

SECONDARY OUTCOMES:
CD4+/CD8+ T lymphocytes count | evolution from baseline to week 48
Genotypic test | if virologic failure occurs
Lipid profile: total, HDL-, LDL-cholesterol and triglyceride levels | evolution from baseline to week 48
Administration of lipid-lowering drugs throughout the study | from baseline to week 48
Cardiovascular risk assessed by the SCORE equation | evolution from baseline to week 48
Patient's satisfaction assessed by 2 scales of type Likert | evolution from baseline to week 48
Adverse events related to antiretroviral treatment | from baseline to week 48
Etravirine plasma trough concentration | Week 4

CONTACTS AND LOCATIONS:
Overall Officials: Eugenia Negredo, MD,PhD, Principal Investigator — Fundación FLS de Lucha Contra el Sida, las Enfermedades Infecciosas y la Promoción de la Salud y la Ciencia
Locations (1):
- Germans Trias i Pujol University Hospital, Badalona, Barcelona, Spain

REFERENCES:
- [Derived] Echeverria P, Bonjoch A, Puig J, Molto J, Paredes R, Sirera G, Ornelas A, Perez-Alvarez N, Clotet B, Negredo E. Randomised study to assess the efficacy and safety of once-daily etravirine-based regimen as a switching strategy in HIV-infected patients receiving a protease inhibitor-containing regimen. Etraswitch study. PLoS One. 2014 Feb 4;9(2):e84676. doi: 10.1371/journal.pone.0084676. eCollection 2014. PMID 24503952